CLINICAL TRIAL: NCT02065037
Title: The Impact of Warmed Carbon Dioxide Insufflation During Colonoscopy on Polyp Detection: A Randomized Controlled Trial
Brief Title: The Impact of Warmed Carbon Dioxide Insufflation During Colonoscopy on Polyp Detection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: CO2 temperature delivered revealed that warmed CO2 was not being delivered.
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Lawrence Hookey, Assistant Professor and Director of Endoscopy, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 6011440; DMED-1658-13 (Other: Queen's University)
Record Dates: First submitted 2014-02-10; First posted 2014-02-17 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Colonic Polyps; Colonic Neoplasms
Keywords: Insufflation; Carbon Dioxide; Colonic Polyps; Colonoscopy; Randomized Controlled Trial
MeSH Terms: conditions — Colonic Polyps; Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Warmed Carbon Dioxide Insufflation (Experimental): warmed carbon dioxide insufflation used in colonoscopy
  Interventions: Device: warmed carbon dioxide insufflation
- Room Temperature Air Insufflation (Active Comparator): room temperature air insufflation used in colonoscopy
  Interventions: Device: room temperature air insufflation

INTERVENTIONS:
Device: room temperature air insufflation — control arm
  Arms: Room Temperature Air Insufflation
Device: warmed carbon dioxide insufflation — comparator arm
  Arms: Warmed Carbon Dioxide Insufflation

SUMMARY:
Colorectal cancer is the second most common cancer in the world and the second leading cause of cancer-related mortality. Colorectal cancers arise from precursor adenomatous polyps in a well characterized adenoma to carcinoma progression. The removal of such precursor lesions reduces colorectal cancer mortality between 30 to 50%. Colonoscopy is used for detection of neoplastic polyps but significant miss rates of such lesions are reported. Methods to reduce spasm of the colon have been investigated to increase adenoma detection rates including the use of warm water irrigation and hyoscine butyl bromide. Carbon dioxide warmed to body temperature is postulated to have spasmolytic effects. Administration of warmed carbon dioxide during colonoscopy may improve polyp detection.

Objective: In this study, colonoscopy using warmed carbon dioxide insufflation will be compared to standard room temperature air insufflation to see if there is a greater detection of polyps per patient.

Methods: Patients undergoing colonoscopy for screening and surveillance indications will be included and randomized to receive either room temperature room air or warmed carbon dioxide (37 degrees Celsius). Endoscopists and patients will be blinded to the intervention. Data on indication, preparation, sedation, withdrawal time will be recorded. Polyp detection rate will be the primary outcome. Secondary outcomes will include adenoma detection rate and advanced lesion detection rates.

DETAILED DESCRIPTION:
study terminated

ELIGIBILITY:
Inclusion Criteria:

-outpatients undergoing routine screening or surveillance colonoscopy for colorectal cancer and / or polyp surveillance at Hotel Dieu Hospital

Exclusion Criteria:

* patients who have undergone colonic resections
* active inflammatory bowel disease
* hereditary polyposis syndromes
* moderate to severe chronic obstructive pulmonary disease
* obstructive sleep apnea requiring continuous positive airway pressure or biphasic positive airway pressure
* neurologic diagnoses affecting ventilation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2014-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Polyp Detection Rate | time of endoscopy

SECONDARY OUTCOMES:
adenoma detection rate | 2 weeks
advanced lesion per patient detection rate | 2 weeks

OTHER OUTCOMES:
cecal intubation rate | day of colonoscopy
withdrawal time | day of colonoscopy
anesthetic doses | day of colonoscopy
quality of bowel preparation | day of colonoscopy
patient comfort by a validated nurse administered comfort score | day of colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Hookey, MD, Principal Investigator — Queens University
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No